CLINICAL TRIAL: NCT02956941
Title: Effect of Behavior Change Communication About Improved Micronutrient Intake on Nutritional Status and Academic Performance of School Age Children in Meskan District, Gurage Zone, South Ethiopia
Acronym: BCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Tsedeke Wolde, Lecturer, Jimma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4088/08; 4086/2016 (Other: Jimma University)
Record Dates: First submitted 2016-10-28; First posted 2016-11-07 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Child Nutrition Disorders
Keywords: Academic performance; Behaviour change communication; Nutritional status; School children; Ethiopia
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCC on Essential Nutrition and Hygiene Actions (ENHAs) (Experimental): Intervention group will be received 12 months on nutrition behavior change communication using two modes (lecture, and posters).
  Interventions: Behavioral: BCC on Essential Nutrition and Hygiene Actions (ENHAs)
- Control cluster (No Intervention): Control group will receive routine dietary practices.

INTERVENTIONS:
Behavioral: BCC on Essential Nutrition and Hygiene Actions (ENHAs) — The behavioral change communication (BCC) on micronutrient intake messages will be implemented based on Essential Nutrition and Hygiene Actions (ENHAs) on micronutrient deficiencies prevention and control. BCC intervention training workshop will be given to science teachers by principal investigator/ senior health professional in local language. Interventions will be delivered to students by their science teachers under the supervision of principal investigator/ school director for the consecutive three times.
  Arms: BCC on Essential Nutrition and Hygiene Actions (ENHAs)

SUMMARY:
A cluster randomized controlled trial was chosen to exploit the robustness of this design to help ascertain the efficacy of the BCC intervention compared to the routine dietary practice. This protocol was developed according to the guidelines of the Consolidated Standards of Reporting Trials (CONSORT) statement extension for cluster randomized trials.

The present study is aims to evaluate the effect of improving micronutrient intake through behavior change communication intervention on nutritional status and academic performance of school age children. Moreover, it may help to prevent or mitigate malnutrition. However to the best knowledge of the authors, BCC intervention using posters, and lecture for school teachers and students have not yet been empirically tested generally in Ethiopia, specifically in the study area context. The present intervention is unique in combining the use of conventional BCC intervention tools, that is, lecture and posters as reminder for intervention reinforcement.

DETAILED DESCRIPTION:
Background: School age children (SAC) are vulnerable to malnutrition which can have adverse effects on their academic performance at school. Micronutrient deficiency affects as many as two billion people in the world. About 250 million people out of this suffer from deficiencies of iron, vitamin A, zinc and iodine are children. Malnutrition or micronutrient deficiencies lead to lower enrolment and completion rates. A nutrition behavior change strategy provides individuals with the necessary resources, knowledge, skills, motivation and reinforcement needed to encourage positive change in health behavior. So far, there are no any studies in the context of the study area in particular and in the country in general on the effect of behavior change communication (BCC) on improving the nutritional status, micronutrient intake and academic performance of school age children.

Objective: The aim of this study protocol is to evaluate the effects of the behavior change communication (BCC) on nutritional status and academic performance of school age children in South Ethiopia. The hypotheses are that the children in the intervention arm will increase their academic performance and improve their nutritional status and micronutrient intake more than the children in the control arm.

Methods: A cluster randomized controlled trial will be carried out to achieve the above mentioned objectives, so that the findings will be used as an input for policies and strategies that will be designed to mitigate the problem. A twelve-month cluster randomized control trial will be conducted in 8 schools of 370 students with ten to fifteen years old. The school intervention will be included BCC for students and science teachers on essential nutrition and hygiene actions (ENHAs) will be provided by background of Health education with Nutritionist. Demographic characteristics, knowledge, attitude & practices (KAP) of micronutrient deficiencies prevention, micronutrient intake, anthropometric measurements (height & weight), and academic performance assessment will be during baseline, mid line and end line assessment. The academic performance of children will be assessed by using end term semester results obtain for English and Mathematics subjects and for the overall subject average.

The trial (n= 376) have two randomly assigned arms: a control cluster schools (CC) and intervention cluster schools (IC) according to their cluster. The IC will be received 12 months on nutrition behavior change communication intervention using two modes (lecture, and posters) while CC receive routine dietary practices. The primary outcomes of this study are stunting, micronutrient intake, dietary diversity score, and academic performance of the children; assess using questionnaires, KAP of micronutrient deficiencies prevention, and anthropometry measurements. Secondary outcomes include thinness, underweight, overweight and obesity.

A multivariate logistic regression analysis will be used to identify independent predictors of nutritional status and academic performance of school age children after controlling for confounding variables. The effect of BCC on nutritional status and academic performance will be determined using generalized estimating equations (GEE) and or linear mixed effects models.

For each of the primary outcomes, stunting, micronutrient intake, dietary diversity score, and academic performance of children, the difference in mean change at follow-up between intervention and control arms will be compared. The hypotheses will be tested under the intent-to-treat principle using Generalized Linear Mixed Models (GLMMs) that will account for the correlation induced by the clustering of children within schools. To further explore the effect of the intervention, GLMMs will be fit that (1) adjust for baseline covariates of interest, consider a priori, relevant to change in nutritional status, KAP of micronutrient deficiencies prevention, micronutrient intake and dietary diversity score; (2) adjust for baseline variables distribute differently between intervention groups; (3) test interaction terms between treatment group and other covariates; and (4) examine completers only. Differences in the secondary outcomes, underweight and obesity will be analyzed in a parallel fashion. Mediating and moderating effects of the factors mentioned above will also be explored.

Discussion: Results of the trial will provide evidence of the effectiveness of the nutrition BCC innovation in school settings of Meskan district. They will provide recommendations for strengthening the nutrition component of behavior change communication in child health services.

ELIGIBILITY:
Participant inclusion criteria:

* All consenting students of classes in all clusters will be recruited for the study.

Participant exclusion criteria:

* School directors and students who are not able to provide informed consent will be ineligible to take part in the trial.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 376 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Linear growth as assessed by mean change in height for age z score | at 6 months (mid line) and at 12 months (end line) of the intervention
  The primary outcome of the study will be linear growth (stunting) as assessed by mean change in height for age z score at 10-15 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
It depends on the data quality and quantity.